CLINICAL TRIAL: NCT03228472
Title: Noninvasive Brain Stimulation Training to Help Recover Brain-related Symptoms
Brief Title: Noninvasive Brain Stimulation Training
Acronym: TrainingNIBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Mario Stampanoni Bassi, Principal Investigator, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRCCS_Neuromed
Record Dates: First submitted 2017-07-13; First posted 2017-07-25 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Patients will undergo a cerebral pacing program listed below and differentiated according to the type of symptom presented. All conventional therapies taken by patients will be recorded by the operators. Patients will be divided into Stimulation and Sham (control) groups and will be evaluated at zero time before starting treatment (T-0W) after 6 weeks to evaluate the effects at the end of treatment (T-6W) and at 12 weeks (T-12W) to evaluate the maintenance of long-term effects. Randomization will be balanced in accordance with age, sex and schooling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Experimental): Cranial - electrical or magnetic stimulation. Stimulation will be different according to clinical conditions, as specified elsewhere.
  Interventions: Device: non invasive brain stimulation
- sham stimulation (Placebo Comparator): Patients will be treated as in the "Real stimulation" arm, but no electrical or magnetic stimulation will be induced.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: non invasive brain stimulation — TDCS stimulation will be administered for 5 consecutive days at 2 mA for 20 minutes.
  TMS stimulation parameters will be: 10 Hz frequency; 100% RMT intensity; Train duration 10 sec (100 stimuli); Inter-train interval 1 minute; n. Total of the terrors 12; Duration of a session about 13 minutes.
  Arms: real stimulation
Device: sham stimulation — Placebo treatment
  Arms: sham stimulation

SUMMARY:
Non-invasive cerebral stimulation techniques have shown potential in the treatment of neurological disorders such as chronic pain, Parkinson's disease, neglect, aphasia, memory, engine deficit and epilepsy In general, non-invasive cerebral stimulation techniques have been shown to be able to induce changes in cortical plasticity that may last even beyond the end of the stimulation period. Considering this potential, there is growing interest in the application of these therapeutic techniques.

Hypotheses Based on these assumptions, the underlying hypothesis behind this project is that the therapeutic use of cranial - electrical or magnetic stimulation - can aid the recovery of various brain injury symptoms.

Specific objectives This study aims to provide preliminary data about the benefits of using cortical stimulation to recover various brain injury symptoms. This will be made possible thanks to the specific skills of a multidisciplinary team of neurologists and physiatrists, healthcare professionals such as physiotherapists, occupational therapists, psychologists, speech therapists and the support of a biomedical engineer. These professional figures are already available at the UCK Neurosurgery of the IRCCS Neuromed directed by the proposer and actively collaborate to optimize the therapeutic exercise of patients with neurological damage.

DETAILED DESCRIPTION:
Introduction TMS is a non-invasive neuronal stimulation of surface areas of the brain that since its introduction in 1985 has been frequently used in neurology as a diagnostic and research tool. TMS uses magnetic fields to induce electrical currents that cross the nervous tissue depolarizing neurons, and reproduced motions generated are recorded as electromyograph potentials. TMS is able to explore the functionality of the cortical-spinal system, measure cortical excitability, mapcortical features, and evaluate brain modulators.

Repetitive transcranial magnetic stimulation (rTMS) is frequently used in the experimental field for cortical function scans and modulation of the intrinsic cortical plasticity. In particular, high frequency rTMS has facilitating effects on cortico-spinal excitability and the low-frequency one is usually inhibitory. rTMS is a method of extreme interest for the possible therapeutic role in conditions of altered cerebral excitability, both psychiatric (schizophrenia, posttraumatic stress disorder, obsessive-compulsive disorder, major depression) and neurological (epilepsy , stroke, degenerative diseases). At experimental level, the actual stimulation is compared with an inactive stimulus called sham, which acts as a control condition.

Direct Transcranial Electric Stimulation (tDCS) requires the application of weak electrical currents directly to the head for several minutes. These currents generate an electric field modulating neural activity based on the application mode. tDCS alters the rate of discharge of neurons. In fact, cathodic polarization applied to the motor cortex can induce a robust reduction in cortical excitability, while anodic polarization increases the excitability of the motor cortex. The short-term effects of tDCS are probably due to a change in neural membrane polarization. Similarly to rTMS, these changes last even after the end of stimulation for periods ranging from minutes to hours. Thus, tDCS can modify performance in many cognitive tasks.

Non-invasive cerebral stimulation have demonstrated a potential for the treatment of neurological disorders such as chronic pain, Parkinson's disease, neglect, aphasia, memory, motor deficiency and epilepsy. In general, non-invasive brain stimulation techniques have shown to induce changes in cortical plasticity that may last even beyond the end of the stimulation period. Considering this potential, there is an increasing interest in the application of these techniques in the therapeutic field.

In our study, we suggest evaluating any variations in the muscular tone of the lower limbs as a result of high frequency repetitive transcranial magnetic stimulation (rTMS) in patients with multiple sclerosis with relapsing-remitting pattern without evidence of medullary demyelination areas. rTMS allows modulation of intracortical excitability and can therefore modify the control of spinal excitability.

Sensory disorders are frequently observed within neurological disorders and are a possible cause of disability. Recent studies based on non-invasive stimulation techniques have shown interesting results in modulation of tactile sensory functions in healthy subjects. tDCS is capable of inducing a plastic change in motor and somatosensory areas. Several studies have reported anodic tDCS stimulation that can reduce both chronic and acute pain in different conditions. In addition, anodic tDCS stimulation can improve the loss of tactile sensitivity resulting from Multiple Sclerosis.

Most patients with Parkinson's Disease develop after several years of treatment with a number of clinical complications, including dyskinesias, involuntary pathological, sometimes frankly, dystonic movements. Pathological Long Term Potentiation (LTP) phenomena were observed in the stigma of parkinsonian rats that developed dyskinesias following L-dopa treatment. Low-frequency electric stimulation of single cells induces a reversal of enhanced synaptic responses, a phenomenon known as depotentiation.

Several authors have observed that in patients with focal dystonia there is a lack of intracortical inhibition of controls. A pilot study examined the effects of slow rTMS on the motor cortex, highlighting normalization of intracortical inhibition and improving clinical symptoms.

The role of TMS in the treatment of major drug-resistant depression has been amply defined. Some early studies demonstrated that a high-frequency focal pacing of the left-sided prefrontal cortex (DLPFC) induced symptom improvement, quantifiable as a reduction in the score to the Hamilton Depression Rating Scale, probably via an increase in the content of brain monoamines. Studies on cerebral blood flow have also shown an increase in activity in the stimulated DLPFC.

It is now accepted that rTMS has the same efficacy, in the most potent drug-resistant depression, of electroconvulsive therapy, with virtually null side effects.

Hypothesis Based on these assumptions, the underlying hypothesis behind this project is that the therapeutic use of cranial - electrical or magnetic stimulation - can aid the recovery of various brain injury symptoms.

Specific objectives This study aims to provide preliminary data about the benefits of using cortical stimulation to recover various brain injury symptoms. This will be made possible thanks to the specific skills of a multidisciplinary team of neurologists and physiatrists, healthcare professionals such as physiotherapists, occupational therapists, psychologists, speech therapists and the support of a biomedical engineer. These professional figures are already available at the UCK Neurosurgery of the IRCCS Neuromed directed by the proposer and actively collaborate to optimize the therapeutic exercise of patients with neurological damage.

Population of the study The sample estimate was made by analogy after a literature analysis. Considering the risk of abandonment quite high, our intention is to recruit at least 100 subjects in a population of patients with cerebral injury who are involved in the neurological department of IRCCS. Neuromed in Pozzilli, featuring the symptoms described below in the inclusion criteria Inclusion and exclusion criteria are specified below.

Experimental design Double-blind prospective study, between randomized, placebo-controlled parallel groups.

Patients will undergo a cerebral pacing program listed below and differentiated according to the type of symptom presented. All conventional therapies taken by patients will be recorded by the operators. Patients will be divided into Stimulation and Sham (control) groups and will be evaluated at zero time before starting treatment (T-0W) after 6 weeks to evaluate the effects at the end of treatment (T-6W) and at 12 weeks (T-12W) to evaluate the maintenance of long-term effects. Randomization will be balanced in accordance with age, sex and schooling.

The physiotherapy or speech therapy approach will be different between patients considering the different types of brain damage and the different levels of disability, according to the rehabilitation unit team for each case.

Spasticity Patients will be evaluated clinically, using a clinical scale to quantify muscle tone in the various districts (Ashworth scale) and neurophysiologically by eliciting the H reflection. The electrophysiological parameters detected will be: M response, H reflex and its M / H ratio. Patients with spasticity to lower limbs will be enrolled in continuous interferon therapy and free of cortisone for at least 30 days.

The runtime rTMS will be applied to the motor at rest (RMT) on the primary motor area for the lower limb, 5 Hz (excitatory) with 20 trains of 10 sec (50 train stimuli, 1000 total stimuli) with intertree intervals of 30 seconds (total 22 min. Ca) on the primary motor cortex for the lower limb and we will measure the H reflex before and after the stimulation session. The treatment will last 2 weeks with daily sessions.

Dyskinesia Patients with clinically diagnosed discontinuous L-Dopa treatment history will be enrolled.

They will be given rTMS for 7 consecutive days with the following stimulation parameters: 1 Hz frequency; 90% Active Motor Threshold intensity; Train duration 899 sec (900 stimuli). At the end of each individual stimulation session patients will be subjected to neurological evaluation of the symptoms.

Sensory Deficits Patients with reduced tactile sensitivity to upper or lower limbs will be enrolled. Patients with peripheral neuropathy, psychiatric disorders, cognitive deficits, epilepsy will be excluded. TDCS stimulation will be administered for 5 consecutive days at 2 mA for 20 minutes. The anode will be placed 2 cm behind the C3 / C4 points of the defective hemisphere. The reference electrode will be positioned over the contralateral control region. Sham stimulation will have the same parameters. Clinical evaluation will be performed before and after treatment, and at a distance of 1, 2 and 4 weeks.

Pain Patients with neuropathic pain in the upper or lower limbs, VAS score of at least 40, will be enrolled in the absence of analgesic treatment for at least one month. Subjects with peripheral neuropathic pain, headache, psychiatric disorders, cognitive deficits, epilepsy will be excluded. TDCS stimulation will be administered as above. The anode will be positioned 2 cm behind the CP's defective hemisphere points. The reference electrode will be positioned over the contralateral control region. Clinical evaluation will be performed before and after treatment, and at a distance of 1, 2 and 4 weeks.

Aphasia Patients with flu-like and non-fluent language disorders will be enrolled, evaluated by clinical scales and clinical visits. TDCS stimulation will be administered for 5 consecutive days, followed by 2 days of pause and subsequent 5 days of 1 mA stimulation for 20 minutes. The anode will be located at the Broca or Wernicke area level. The cathode will be placed on the homologous counterpartical area of the anode. Logopedic therapy will be coupled to true tDCS stimulation and sham. Clinical evaluation will be performed before and after treatment, and at a distance of 1, 2 and 4 weeks.

Dysphagia Patients with swallowing disorders will be enrolled, evaluated by clinical scales, logopedic visit, Otorhinolaryngology visit. TDCS stimulation will be administered for 5 consecutive days at 2 mA for 20 minutes. The anode will be positioned at the level of the dominant motor cortex to control the muscles of the swallowing. The reference electrode will be positioned over the contralateral control region. Logopedic therapy will be coupled to true tDCS stimulation and sham. Clinical evaluation will be performed before and after treatment, and at a distance of 1, 2 and 4 weeks by logopedic, neurophysiological and ORL assessment.

Major Depression In the study, 15 patients with major DSM-IV depression diagnosed with proven drug resistance will be enrolled. Of these, five will be submitted to rTMS of the left dorsolateral prefrontal cortex (DLPFC), five at rTMS of the right DLPFC and five at sham stimulation. The study will be conducted in single blind. The rTMS session will last (15) consecutive days. The stimulation parameters will be: 10 Hz frequency; 100% RMT intensity; Train duration 10 sec (100 stimuli); Inter-train interval 1 minute; n. Total of the terrors 12; Duration of a session about 13 minutes. Hamilton Depression Rating Scale will be administered on the first day before stimulation, and on the last day after stimulation.

Expected results The present study aims to provide preliminary data on the benefits of cortical stimulation for the recovery of various brain injury symptoms.

The expected result is that neurostimulation training potentiates the recovery of the various symptoms considered in the present study, resulting in brain damage.

ELIGIBILITY:
The sample estimate was made by analogy after a literature analysis. Considering the risk of abandonment quite high, our intention is to recruit at least 100 subjects in a population of patients with cerebral injury who are involved in the neurological department of I.R.R.C.S. Neuromed by Pozzilli, featuring the symptoms described below in the inclusion criteria

Inclusion criteria:

* Males or females aged between 18 and 80;
* Presence of: Disinfection, Multiple Sclerosis, Depression, Sensory Disorder or Neuropathic Pain;
* Female subjects can not be pregnant, can not breastfeed, have been born at least three months before the beginning of the study, undertake not to schedule a pregnancy for the duration of the study;
* Patients should be able to follow protocol guidelines throughout the study;
* Patients should be able to understand the aims and risks of the study;
* Signature of informed consent, approved by our Ethics Committee.

Exclusion criteria:

* Tumors or systemic infections;
* Patients with impaired hepatic function (ALT> 3 x Upper Limit Normal (ULN), Alkaline Phosphatase> 2 x ULN, bilirubin tot> 2 x ULN if associated with any increase in ALT or alkaline phosphatase); Severe or moderate renal failure;
* Patients with TMS or tDCS (pacemaker, intracerebral metal clip, epilepsy ...)
* Patients with other pathologies which, according to the scientific officer's opinion, prevent recruitment;
* Patients unable to even partially understand and want.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Barthel's Activities of Daily Living (ADL) (O'Sullivan et al 2007) | up to 3 years
  Abilities of daily living
FIM | up to 3 years
  Functional Independence Measurement (FIM) (Chumney et al., 2010)
stroke | up to 3 years
  NIH Stroke Scale / Score (NIHSS)
disability | up to 3 years
  Expanded Disability Status Scale (EDSS) (Kurtzke, 1983)
parkinson | up to 3 years
  Unified Parkinson's Disease Rating Scale (Rammer et al. )
depression | up to 3 years
  Beck Depression Inventory (BDI) (Beck, 1972)

SECONDARY OUTCOMES:
neuronal plasticity | up to 3 years
  Transcranial Magnetic Stimulation (TMS) will be used to evaluate the change of neuronal plasticity in a subgroup of patients who will not present contraindications to the method. The TMS uses short-lived magnetic fields and high intensity applied at the scalp level to activate the neurons of a small region of the cerebral cortex through an electromagnetic induction. When these impulses are applied repeatedly, it is possible to induce plastic modification of cortical excitability. If these changes are induced at the level of the motor cortex, they can be measured by recording a motor evoked potential (MEP) at the muscle level represented at the stimulated region level. Any increase or decrease in AMP amplitude, which persists after the end of TMS repetitive stimulation, indicates that there have been changes in the cortical, LTP or depression (LTD).
posture | up to 3 years
  Stabilometric Platform
locomotion | up to 3 years
  Gait Analysis
deglutition | up to 3 years
  Electrophysiological and Fiberendoscopic Deglutition Study
Cognition | up to 3 years
  ad-hoc task

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, MD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antal A, Brepohl N, Poreisz C, Boros K, Csifcsak G, Paulus W. Transcranial direct current stimulation over somatosensory cortex decreases experimentally induced acute pain perception. Clin J Pain. 2008 Jan;24(1):56-63. doi: 10.1097/AJP.0b013e318157233b. PMID 18180638
- [Background] Barker AT, Jalinous R, Freeston IL. Non-invasive magnetic stimulation of human motor cortex. Lancet. 1985 May 11;1(8437):1106-7. doi: 10.1016/s0140-6736(85)92413-4. No abstract available. PMID 2860322
- [Background] Baxter LR Jr. Neuroimaging studies of obsessive compulsive disorder. Psychiatr Clin North Am. 1992 Dec;15(4):871-84. PMID 1461802
- [Background] Ben-Shachar D, Belmaker RH, Grisaru N, Klein E. Transcranial magnetic stimulation induces alterations in brain monoamines. J Neural Transm (Vienna). 1997;104(2-3):191-7. doi: 10.1007/BF01273180. PMID 9203081
- [Background] Boggio PS, Zaghi S, Lopes M, Fregni F. Modulatory effects of anodal transcranial direct current stimulation on perception and pain thresholds in healthy volunteers. Eur J Neurol. 2008 Oct;15(10):1124-30. doi: 10.1111/j.1468-1331.2008.02270.x. Epub 2008 Aug 20. PMID 18717717
- [Background] Chen R, Classen J, Gerloff C, Celnik P, Wassermann EM, Hallett M, Cohen LG. Depression of motor cortex excitability by low-frequency transcranial magnetic stimulation. Neurology. 1997 May;48(5):1398-403. doi: 10.1212/wnl.48.5.1398. PMID 9153480
- [Background] Dieckhofer A, Waberski TD, Nitsche M, Paulus W, Buchner H, Gobbele R. Transcranial direct current stimulation applied over the somatosensory cortex - differential effect on low and high frequency SEPs. Clin Neurophysiol. 2006 Oct;117(10):2221-7. doi: 10.1016/j.clinph.2006.07.136. Epub 2006 Aug 23. PMID 16931142
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Greenberg BD, George MS, Martin JD, Benjamin J, Schlaepfer TE, Altemus M, Wassermann EM, Post RM, Murphy DL. Effect of prefrontal repetitive transcranial magnetic stimulation in obsessive-compulsive disorder: a preliminary study. Am J Psychiatry. 1997 Jun;154(6):867-9. doi: 10.1176/ajp.154.6.867. PMID 9167520
- [Background] Hamdy S, Rothwell JC. Gut feelings about recovery after stroke: the organization and reorganization of human swallowing motor cortex. Trends Neurosci. 1998 Jul;21(7):278-82. doi: 10.1016/s0166-2236(97)01212-5. PMID 9683316
- [Background] Hummel F, Celnik P, Giraux P, Floel A, Wu WH, Gerloff C, Cohen LG. Effects of non-invasive cortical stimulation on skilled motor function in chronic stroke. Brain. 2005 Mar;128(Pt 3):490-9. doi: 10.1093/brain/awh369. Epub 2005 Jan 5. PMID 15634731
- [Background] Hummel F, Cohen LG. Improvement of motor function with noninvasive cortical stimulation in a patient with chronic stroke. Neurorehabil Neural Repair. 2005 Mar;19(1):14-9. doi: 10.1177/1545968304272698. PMID 15673839
- [Background] Matsunaga K, Nitsche MA, Tsuji S, Rothwell JC. Effect of transcranial DC sensorimotor cortex stimulation on somatosensory evoked potentials in humans. Clin Neurophysiol. 2004 Feb;115(2):456-60. doi: 10.1016/s1388-2457(03)00362-6. PMID 14744588
- [Background] Mori F, Codeca C, Kusayanagi H, Monteleone F, Buttari F, Fiore S, Bernardi G, Koch G, Centonze D. Effects of anodal transcranial direct current stimulation on chronic neuropathic pain in patients with multiple sclerosis. J Pain. 2010 May;11(5):436-42. doi: 10.1016/j.jpain.2009.08.011. Epub 2009 Dec 16. PMID 20018567
- [Background] Mori F, Nicoletti CG, Kusayanagi H, Foti C, Restivo DA, Marciani MG, Centonze D. Transcranial direct current stimulation ameliorates tactile sensory deficit in multiple sclerosis. Brain Stimul. 2013 Jul;6(4):654-9. doi: 10.1016/j.brs.2012.10.003. Epub 2012 Oct 27. PMID 23122918
- [Background] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Background] Pridmore S. Substitution of rapid transcranial magnetic stimulation treatments for electroconvulsive therapy treatments in a course of electroconvulsive therapy. Depress Anxiety. 2000;12(3):118-23. doi: 10.1002/1520-6394(2000)12:33.0.CO;2-G. PMID 11126185
- [Background] Que M, Schiene K, Witte OW, Zilles K. Widespread up-regulation of N-methyl-D-aspartate receptors after focal photothrombotic lesion in rat brain. Neurosci Lett. 1999 Oct 1;273(2):77-80. doi: 10.1016/s0304-3940(99)00598-4. PMID 10505620
- [Background] Ragert P, Dinse HR, Pleger B, Wilimzig C, Frombach E, Schwenkreis P, Tegenthoff M. Combination of 5 Hz repetitive transcranial magnetic stimulation (rTMS) and tactile coactivation boosts tactile discrimination in humans. Neurosci Lett. 2003 Sep 11;348(2):105-8. doi: 10.1016/s0304-3940(03)00745-6. PMID 12902029
- [Background] Ragert P, Franzkowiak S, Schwenkreis P, Tegenthoff M, Dinse HR. Improvement of tactile perception and enhancement of cortical excitability through intermittent theta burst rTMS over human primary somatosensory cortex. Exp Brain Res. 2008 Jan;184(1):1-11. doi: 10.1007/s00221-007-1073-2. Epub 2007 Aug 7. PMID 17680239
- [Background] Ragert P, Vandermeeren Y, Camus M, Cohen LG. Improvement of spatial tactile acuity by transcranial direct current stimulation. Clin Neurophysiol. 2008 Apr;119(4):805-11. doi: 10.1016/j.clinph.2007.12.001. Epub 2008 Jan 18. PMID 18203660
- [Background] Ridding MC, Sheean G, Rothwell JC, Inzelberg R, Kujirai T. Changes in the balance between motor cortical excitation and inhibition in focal, task specific dystonia. J Neurol Neurosurg Psychiatry. 1995 Nov;59(5):493-8. doi: 10.1136/jnnp.59.5.493. PMID 8530933
- [Background] Rogalewski A, Breitenstein C, Nitsche MA, Paulus W, Knecht S. Transcranial direct current stimulation disrupts tactile perception. Eur J Neurosci. 2004 Jul;20(1):313-6. doi: 10.1111/j.0953-816X.2004.03450.x. PMID 15245504
- [Background] Rossini PM, Calautti C, Pauri F, Baron JC. Post-stroke plastic reorganisation in the adult brain. Lancet Neurol. 2003 Aug;2(8):493-502. doi: 10.1016/s1474-4422(03)00485-x. PMID 12878437
- [Background] Siebner HR, Tormos JM, Ceballos-Baumann AO, Auer C, Catala MD, Conrad B, Pascual-Leone A. Low-frequency repetitive transcranial magnetic stimulation of the motor cortex in writer's cramp. Neurology. 1999 Feb;52(3):529-37. doi: 10.1212/wnl.52.3.529. PMID 10025782
- [Background] Siebner HR, Rothwell J. Transcranial magnetic stimulation: new insights into representational cortical plasticity. Exp Brain Res. 2003 Jan;148(1):1-16. doi: 10.1007/s00221-002-1234-2. Epub 2002 Nov 5. PMID 12478392
- [Background] Speer AM, Kimbrell TA, Wassermann EM, D Repella J, Willis MW, Herscovitch P, Post RM. Opposite effects of high and low frequency rTMS on regional brain activity in depressed patients. Biol Psychiatry. 2000 Dec 15;48(12):1133-41. doi: 10.1016/s0006-3223(00)01065-9. PMID 11137053
- [Background] Tegenthoff M, Ragert P, Pleger B, Schwenkreis P, Forster AF, Nicolas V, Dinse HR. Improvement of tactile discrimination performance and enlargement of cortical somatosensory maps after 5 Hz rTMS. PLoS Biol. 2005 Nov;3(11):e362. doi: 10.1371/journal.pbio.0030362. Epub 2005 Oct 18. PMID 16218766
- [Background] Wassermann EM, Grafman J, Berry C, Hollnagel C, Wild K, Clark K, Hallett M. Use and safety of a new repetitive transcranial magnetic stimulator. Electroencephalogr Clin Neurophysiol. 1996 Oct;101(5):412-7. PMID 8913194